CLINICAL TRIAL: NCT00761618
Title: Effectiveness of Daily Versus Three Times a Week Drainage After Placement of Intrapleural Catheters for the Palliative Management of Pleural Effusions Associated With Malignancies
Brief Title: Intrapleural Catheter Daily Versus Three Times a Week Drainage
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0808; NCI-2012-01673 (Registry Identifier: NCI CTRP-Clinical Trials Reporting Registry)
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Advanced Cancer; Pleural Effusion
Keywords: Intrapleural catheter; IPC; Pleurodesis; PD; Pleural effusion; Fluid in the chest cavity; Recurrent malignant pleural effusion; MPE; Pleural inflammatory response
MeSH Terms: conditions — Pleural Effusion; Pleural Effusion, Malignant | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Daily (Experimental): Intrapleural Catheters (IPC) drained every day
  Interventions: Procedure: Intrapleural catheter (IPC) drained; Procedure: IPC Placement; Radiation: Chest X-Ray
- Arm 2 - 3 Times a Week (Experimental): IPC drained 3 times a week
  Interventions: Procedure: Intrapleural catheter (IPC) drained; Procedure: IPC Placement; Radiation: Chest X-Ray

INTERVENTIONS:
Procedure: Intrapleural catheter (IPC) drained — IPC drained daily (Group 1) or 3 times per week (Group 2)
Procedure: IPC Placement — IPC placed in chest cavity to drain excess fluid
  Other Names: Indwelling Pleural Catheter
Radiation: Chest X-Ray — Chest X-Rays at 3 and 6 month follow up visits

SUMMARY:
The goal of this clinical research study is to learn if draining the IPC every day is better at than draining it 3 times a week.

DETAILED DESCRIPTION:
An IPC is a silicone (rubberlike) tube that is inserted into the chest cavity to drain excess fluid that is in your chest. At MD Anderson, patients are told to drain their IPC every day. At other institutions, patients are told to drain their IPC less often.

Before IPC Placement:

Before you can have the IPC inserted, the following tests and procedures will be performed to help the doctor decide if you need to have an IPC inserted:

* You will perform a 6 minute walk test to learn your check your breathing ability and fatigue level. To perform the walk test, you will be asked to walk as far as possible around cones on a flat indoor course that is about 40 yards long. You will walk at your own pace and can take breaks at any time if necessary.
* After signing this consent, you will fill out 2 questionnaires asking questions about how you feel and any symptoms you may have. These questionnaires will take about 20-30 minutes to complete.

IPC placement:

You will have an IPC placed to drain the fluid in your chest cavity. You will be given a separate consent for to sign for this procedure and your doctor will give you detailed instructions regarding the procedure itself.

Study Groups:

A chest x-ray will be performed right after the IPC placement. You will be randomly assigned (as in the flip of a coin) to 1 of 2 groups, after your chest x-ray or the following day when you return to clinic for follow up. Group 1 will have their IPC drained every day, and Group 2 will have their IPC drained 3 times a week (Monday, Wednesday, and Friday or Tuesday, Thursday, and Saturday). You will be given detailed instructions on when and how to drain your catheter.

Follow-Up Visits:

Two (2) weeks after you receive the IPC, you will return to the clinic for a follow-up visit so the doctor can check your IPC for possible leaking, infection, and see how much pleural fluid has drained. After the follow-up visit at 2 weeks, you will come into the clinic every 4 weeks until your IPC is removed. During each follow-up visit the following tests and procedures will be performed to see how your condition has changed:

* You will have a chest x-ray to see if the amount of pleural fluid has decreased and to see if your lung has re-expanded.
* You will perform the 6 minute walk test.
* You will complete the same 2 questionnaires.
* The IPC will be drained.

After the IPC is removed, at 3 and 6 months, you will have follow-up visits at M. D. Anderson or at your local doctor's office. At these visits you will have chest x-rays to see if the pleural fluid has come back or not.

The study personnel will contact you by phone, email or mail periodically during the study and at 3 months and 6 months after the IPC has been removed to check on your status. The phone calls, email, or mail follow-up will take about 5-10 minutes to complete. You will be asked how you are doing and if you have any questions or concerns that you may want to discuss with the your doctor. You will also be asked if you have had a chest x-ray since being off study. If you have had an x-ray, you will be asked to share the results with the study doctor.

This is an investigational study.

Up to 250 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic pleural effusion requiring placement of an IPC.
2. Signed informed consent prior to any study related procedures.
3. Subject must be age 18 years or over.

Exclusion Criteria:

1. Any of the following interventions on the affected hemithorax: prior IPC, prior chest tube placement, history of chemical or mechanical pleurodesis, history of thoracotomy within 4 weeks incompletely healed surgical incision before randomization.
2. Evidence of empyema or history of empyema of the affected hemithorax
3. Non-correctable bleeding diathesis
4. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
5. Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the Principal Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol.
6. Participation in any clinical trial that prevents randomization of the subject to either strategy.
7. Clinical evidence of skin infection at the potential site of IPC placement.
8. Current or prior IPC placement, or any intervention to manage recurrent malignant pleural effusion on the contralateral hemithorax (excluding thoracentesis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2008-08-22 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Time to Pleurodesis (TTP) | 2 weeks after intrapleural catheter placement
  Time to pleurodesis (TTP), defined as the time from catheter insertion to catheter removal.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A. Jimenez, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org